CLINICAL TRIAL: NCT00998582
Title: Artery Elasticity After Switch From Epzicom to Truvada
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Low enrollment
Sponsor: Hennepin Healthcare Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PCC-004
Record Dates: First submitted 2009-10-19; First posted 2009-10-20 (Estimated); Results first posted 2012-03-23 (Estimated); Last update posted 2012-10-08 (Estimated); Status verified 2012-10

CONDITIONS: HIV Infections
Keywords: Cardiovascular Disease; HIV Infection; Abacavir; Artery Elasticity; Treatment experienced
MeSH Terms: conditions — HIV Infections; Cardiovascular Diseases | interventions — Tenofovir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Abacavir (Active Comparator): Participants randomized to this arm will continue abacavir and their other HIV medications with no changes
  Interventions: Drug: Tenofovir disoproxil
- Tenofovir (Experimental): Participants randomized to this arm will switch from taking abacavir (co-formulated with lamivudine as Epzicom) and start taking tenofovir (co-formulated with emtricitabine as Truvada), and continue their other HIV medications
  Interventions: Drug: Tenofovir disoproxil

INTERVENTIONS:
Drug: Tenofovir disoproxil — Participants taking an abacavir-based HIV treatment regimen will be randomized to switch to a tenofovir-based regimen or continue taking abacavir.

SUMMARY:
Recent research as suggested that use of the HIV medication abacavir (Ziagen, or co-formulated with lamivudine as Epzicom) may increase risk for heart disease, though findings from multiple studies have been inconsistent. This pilot study will examine vascular function, a marker of heart disease risk, among patients taking abacavir as part of their HIV medications and are then randomized to: 1) switch to tenofovir, another HIV medication, or 2) continue to take abacavir.

ELIGIBILITY:
Inclusion Criteria:

* Adult (≥18 years) males or non-pregnant females, non-lactating females.
* HIV-infected participants currently receiving fixed-dose abacavir/lamivudine based regimen for ≥3 months preceding the screening visit.
* HIV-infection documented by a positive HIV-1 antibody (confirmatory western-blot) or an HIV RNA level ≥1000 copies/mL
* Two consecutive plasma HIV RNA concentrations below the limit of detection for clinical-based assays used for HCMC and ANW HIV clinics. The 1st HIV RNA concentration must be at least 3 months prior to study entry.
* Subjects receiving lipid lowering agents will be allowed; however, dosing for these medications must be stable for ≥3 months prior to study entry
* Adequate renal function defined as a calculated creatinine clearance (CLCr) ≥50 mL/min according to the Cockcroft-Gault formula:

  * MALE: (140 - age in years) x (wt in kg) = CLCr (mL/min) 72 x (serum creatinine in mg/dL)
  * FEMALE: (140 - age in years) x (wt in kg) x 0.85 = CLCr (mL/min) 72 x (serum creatinine in mg/dL)
* Negative serum pregnancy test (females of childbearing potential only)
* Hepatic transaminases (AST and ALT) ≤ 5 x upper limit of normal (ULN).
* Males and females (of childbearing potential) must agree to avoid pregnancy by sexual abstinence, or utilization of a highly effective method of birth control throughout the study period and for 30 days following discontinuation of study drug (refer to Appendix A for definitions of 'childbearing potential' and 'highly effective method of birth control')

Exclusion Criteria:

* Subjects with known resistance to abacavir, lamivudine, tenofovir DF, or emtricitabine at anytime in the past (including but not limited to K65R, L74V/I, M184V/I, or thymidine analog mutations).
* A new AIDS-defining condition diagnosed (with the exception of CD4 criteria) within 30 days of baseline
* Previous therapy with agents with systemic myelosuppressive, pancreatoxic, hepatotoxic or cytotoxic potential within 3 months of study entry or the expectation for such therapy at the time of enrollment
* Proven or suspected acute hepatitis in the 30 days prior to study entry
* Receiving ongoing therapy with any of the following (administration of any of the following medications must be discontinued at least 30 days prior to the baseline visit and for the duration of the study period):

  * Nephrotoxic agents (aminoglycoside antibiotics, amphotericin B, cidofovir, cisplatin, foscarnet, IV pentamidine, other agents with significant nephrotoxic potential)
  * Adefovir dipivoxil
  * Probenecid
  * Systemic chemotherapeutic agents (i.e., cancer treatment medications)
  * Systemic corticosteroids
  * Interleukin-2 (IL-2)
* Evidence of gastrointestinal malabsorption syndrome or chronic nausea or vomiting which may confer an inability to receive an orally administered medication.
* Current alcohol or substance abuse judged by the investigator to potentially interfere with subject adherence
* Malignancy other than cutaneous Kaposi's sarcoma (KS) or basal cell carcinoma. Participants with biopsy-confirmed cutaneous KS are eligible, but must not have received any systemic therapy for KS within 30 days of baseline and are not anticipated to require systemic therapy during the study.
* Active, serious infections (other than HIV-1 infection) requiring parenteral antimicrobial therapy within 15 days prior to screening.
* Prior history of significant renal or bone disease.
* Any other clinical condition or prior therapy that, in the opinion of the investigator, would make the subject unsuitable for the study or unable to comply with the dosing requirements.
* Known hypersensitivity to the study drugs, the metabolites or formulation excipients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2009-10; Primary Completion 2011-06 (Actual); Study Completion 2011-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jason Baker, MD, MS, Principal Investigator — University of Minnesota; HCMC
Locations (2):
- United States (2):
  - Hennepin County Medical Center, Minneapolis, Minnesota
  - Abbott Northwestern Hospital and Clinics, Minneapolis, Minnesota

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Abacavir | Tenofovir
Started | 13 | 14
Completed | 13 | 14
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Abacavir | Tenofovir | Total
Number analyzed (Participants) | 13 | 14 | 27
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 13 | 14 | 27
  >=65 years | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 47 (7) | 43 (9) | 46 (8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 0 | 1
  Male | 12 | 14 | 26
Region of Enrollment [Number; unit: participants]
  United States | 13 | 14 | 27

OUTCOME MEASURES:

1. Primary Outcome: Change in Small Artery Elasticity (mL/mmHg x100) From Baseline to Week 24
Description: Small artery elasticity is a measure of vascular function, estimated through analysis of the blood pressure waveform. A sensor is placed on wrist over the radial pulse. The blood pressure waveform of the pulse is recorded and analyzed the elasticity, or compliance, of the small (and large) vasculature. Impaired artery elasticity, or increased stiffness, is an early sign of vascular disease that predicts risk for future cardiovascular events.
Time Frame: Change from baseline to 24 weeks
Population: Small artery elasticity was measured at baseline and week 24 in all participants. Outcome was change in small artery elasticity (mL/mmHg x100) from baseline to week 24
Measure: Median (Inter-Quartile Range); unit: ml/mmHg x100
Arm/Group | Abacavir | Tenofovir
Number analyzed (Participants) | 13 | 14
ml/mmHg x100 | 0.2 [-0.5 to 2.3] | -1.3 [-2.8 to 2.7]

2. Primary Outcome: Outcome Was Change in Large Artery Elasticity (mL/mmHg x100) From Baseline to Week 24
Description: Large artery elasticity is a measure of vascular function, estimated through analysis of the blood pressure waveform. A sensor is placed on wrist over the radial pulse. The blood pressure waveform of the pulse is recorded and analyzed the elasticity, or compliance, of the large (and small) vasculature. Impaired artery elasticity, or increased stiffness, is an early sign of vascular disease.
Time Frame: Change from baseline to 24 weeks
Population: Large artery elasticity was measured at baseline and week 24 in all participants. Outcome was change in large artery elasticity (mL/mmHg x10) from baseline to week 24
Measure: Median (Inter-Quartile Range); unit: ml/mmHg x10
Arm/Group | Abacavir | Tenofovir
Number analyzed (Participants) | 13 | 14
ml/mmHg x10 | -0.2 [-1.7 to 3.1] | -0.4 [-1.9 to 1.7]

ADVERSE EVENTS:
Arm/Group | Abacavir | Tenofovir
Serious Adverse Events (participants affected / at risk) | 0/13 | 0/14
Other Adverse Events (participants affected / at risk) | 0/13 | 0/14

LIMITATIONS AND CAVEATS:
Study stopped early due to low/inadequate enrollment and findings are subsequently limited by low power to detect differences.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No